CLINICAL TRIAL: NCT06500156
Title: Metabolic Cluster Analysis in Septic Shock Patients Undergoing Hemodynamic Resuscitation. A Multicenter Observational Study
Brief Title: Metabolic Cluster Analysis in Septic Shock Patients
Acronym: ACMEcat
Status: Recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jaume Mesquida, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 20235121
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Septic Shock
Keywords: septic shock; hemodynamic resuscitation; cardiovascular monitoring
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock: Septic shock patients within the first 24 hours of ICU admission, and selected by the attending physician for performing a fluid challenge (FC) due to suspected tissue hypoperfusion.
  Interventions: Other: Fluid challenge

INTERVENTIONS:
Other: Fluid challenge — Rapid infusion (< 15 minutes) of a fluid bolus of crystalloids (200 to 500cc)

SUMMARY:
Observational study including septic shock patients within 24 hours of ICU admission, monitored with a cardiac output estimation system, with ongoing resuscitation. Hemodynamic and metabolic parameters before and after a fluid challenge (FC) will be measured.

ELIGIBILITY:
Inclusion Criteria:

- Septic shock patients within the first 24 hours of ICU admission, and selected by the attending physician for performing a fluid challenge (FC) due to suspected tissue hypoperfusion (elevated lactate and/or ScvO2 < 70%).

Exclusion Criteria:

* Age under 18 years old
* Uncontrolled hemodynamic instability, defined as the need for significant changes in vasopressor support (> 10% from baseline dose) within the 15-minute period prior to, and/or during the administration of fluids.
* Patients receiving continuous renal replacement therapies, since the CO values obtained from the thermodilution techniques might be potentially affected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic shock patients within the first 24 hours of ICU admission, and selected by the attending physician for performing a fluid challenge (FC) due to suspected tissue hypoperfusion.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
VO2-response | 30 minutes
  Percentage increase in VO2 as results of the fluid challenge

SECONDARY OUTCOMES:
Organ failure | 4 days
  Assessment of the SOFA score at day 1, 2 and 4
Mortality | 28 days
  Mortality within the first 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Parc Taulí, Sabadell, Barcelona, Spain